CLINICAL TRIAL: NCT04771793
Title: Physical Restraint of Critically Ill Patients: Prevalence, Properties and Associated Delirium Score
Brief Title: Physical Restraint of Critically Ill Patients
Status: Completed | Type: Observational
Sponsor: Meir Medical Center (Other)
Responsible Party: Principal Investigator, sara dichtwald, Dr., Meir Medical Center
Other Study IDs: 0420-20-MMC
Record Dates: First submitted 2021-02-02; First posted 2021-02-25 (Actual); Last update posted 2023-03-15 (Actual); Status verified 2023-03

CONDITIONS: Delirium
MeSH Terms: conditions — Delirium

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group A- before implentation of physical restraint protocols
  Interventions: Behavioral: new physical restraint protocols
- Group B- after implentation of physical restraint protocols
  Interventions: Behavioral: new physical restraint protocols

INTERVENTIONS:
Behavioral: new physical restraint protocols — new physical restraint protocols

SUMMARY:
Background: Physical restraint of patients in the intensive care unit (ICU) is a common practice, with estimated prevalence of 50% of all ICU patients, with and without invasive ventilation support(1). The prevalence of physical restraint varies between ICU's according to patient population (surgical, cardiac, trauma, burns and general intensive care patients). In mechanically ventilated patients, the physical restriction (tying the patient) is carried out frequently in addition to pharmacological treatment with analgesic and sedative medications, in order to prevent falling, self-inflicted injury or accidental removal of essential medical devices (tracheobronchial tubes, central venous infusions, drains, etc.) by the patient. In non-ventilated patients, physical restraint is often carried out in patients with delirium or cognitive decline, in addition to pharmacological anti -delirium therapy (1).

However, physical restraint has many drawbacks, including injuries to the skin and the soft tissues, blood vessels, peripheral nerves, muscle and skeleton (2). In addition, physical restraint may exacerbate symptoms of restlessness and delirium and even increase the risk of developing post-traumatic stress disorder in these patients (3,4).

Despite the high prevalence of physical restraint of ICU patients, with its disadvantages and advantages, currently there are no consensual criteria for physical restraint and the decision when and how long to use it is at the discretion of the attending physician. It is important to note that in recent years there has been a tendency to reduce the amount of sedation that mechanically ventilated patients are given, which may lead to an increase in the incidence of physical restraint of patients who are fully or partially conscious (5).

DETAILED DESCRIPTION:
Background: Physical restraint of patients in the intensive care unit (ICU) is a common practice, with estimated prevalence of 50% of all ICU patients, with and without invasive ventilation support(1). The prevalence of physical restraint varies between ICU's according to patient population (surgical, cardiac, trauma, burns and general intensive care patients). In mechanically ventilated patients, the physical restriction (tying the patient) is carried out frequently in addition to pharmacological treatment with analgesic and sedative medications, in order to prevent falling, self-inflicted injury or accidental removal of essential medical devices (tracheobronchial tubes, central venous infusions, drains, etc.) by the patient. In non-ventilated patients, physical restraint is often carried out in patients with delirium or cognitive decline, in addition to pharmacological anti -delirium therapy (1).

However, physical restraint has many drawbacks, including injuries to the skin and the soft tissues, blood vessels, peripheral nerves, muscle and skeleton (2). In addition, physical restraint may exacerbate symptoms of restlessness and delirium and even increase the risk of developing post-traumatic stress disorder in these patients (3,4).

Despite the high prevalence of physical restraint of ICU patients, with its disadvantages and advantages, currently there are no consensual criteria for physical restraint and the decision when and how long to use it is at the discretion of the attending physician. It is important to note that in recent years there has been a tendency to reduce the amount of sedation that mechanically ventilated patients are given, which may lead to an increase in the incidence of physical restraint of patients who are fully or partially conscious (5).

Objectives: In the first stage of our planned study (in this study) - we would like to assess the prevalence of physical restraint in ICU patients, both with and without mechanical ventilation support, their clinical characteristics and the rate of delirium among them. In the second stage of the study (in a future study) - we plan to install specific protocols for physical restraint, aiming to decrease the rate of physical restraint of patients in our ICU.

The data obtained from the first phase of the study can help us characterize the patients who require physical restraint in the ICU, which from we will attempt to generate protocols that will help us reduce the prevalence of physical restraint in the unit. For example, if the group of patients who required physical restraint tended to experience delirium more often, as measured by the RASS score, we could formulate a special protocol for the treatment of delirium in these patients, which might reduce the need for physical restraint in some cases. We can address factors that may alter the incidence of delirium, such as emphasizing the importance of renewing as soon as possible all regular patients' pharmacological therapy with antipsychotic drugs, if any, or to soon start treatment to prevent withdrawal syndrome (in case of chronic ethanol abuse, or regular benzodiazepine treatment. Alternative measures can also be used to decrease delirium prevalence, such as presence of the patient's family member, music, television, maintaining the patient's room dark at night hours, etc.), as well as other measures. The characterization of those patients is essential for the formulation of such treatment protocols.

Methods and materials:

Study type: Retrospective study based on data collection. Data will be extracted from the hospital computerized systems. The study will include all our ICU admitted patients from 1.1.2020 to 31.12.2020. About 1000 patients total.

Inclusion criteria: All patients aged 18--99 admitted to the General Intensive Care Unit from January 2020 to the end of December 2020.

Data collection: Retrospective observational data collection from hospital records and computerized systems (Chameleon system and iMDsoft software).

Collected data: Age, gender, hospital and ICU admission times, ventilation days, 28-day mortality, past medical history including chronic medication therapy, APACHE-2 score, admission lactate level, need for pressor or inotropic support, need for dialysis, need for tracheostomy, type of ICU admission (Infectious, trauma etc.), delirium score measured by the RASS score, need for physical restraint, duration of physical restraint, prevalence of self extubation, prevalence of self-inflicted injuries including falls and inadvertent retrieval of tubes or other medical devices.

Study group size: 1000 patients. Statistical analysis: All demographic and intra-patient parameters will be statistically examined by a qualified statistician depending on the type of data. The current study group will be the control group (before intervention), and the second group will be the treatment group (after intervention, i.e. after creating and installing new physical restraint protocols in the ICU) .We will use the Chi square test to analyze the discrete data and the Mann-Whitney test to analyze the continuous data.

ELIGIBILITY:
Inclusion Criteria: All patients aged 18--99 admitted to the General Intensive Care Unit from January 2020 to December 2020.

-

Exclusion Criteria: None.

-

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients aged 18--99 admitted to the General Intensive Care Unit from January 2020 to December 2020.
Sampling Method: Non-Probability Sample
Enrollment: 992 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2023-03-14 (Actual); Study Completion 2023-03-14 (Actual)

PRIMARY OUTCOMES:
Prevalence of physical restraint in ICU patients | 1 year (January 2020 - December 2020.
  To assess the prevalence of physical restraint in ICU patients (%), both with and without mechanical ventilation support

CONTACTS AND LOCATIONS:
Locations (1):
- Meir medical center Kfar Saba, Kfar Saba, Israel

REFERENCES:
- [Derived] Cohen S, Meyer A, Ifrach N, Dichtwald S. Physical restraint and associated agitation. Nurs Crit Care. 2024 Sep;29(5):1132-1141. doi: 10.1111/nicc.13130. Epub 2024 Jul 14. PMID 39004848